CLINICAL TRIAL: NCT05671718
Title: Bring BPaL2Me Trial Comparing Nurse-Led RR-TB Treatment in Primary Care to Physician-Led, Hospital-Based Outpatient RR-TB Treatment: A Cluster Randomized, Non-Inferiority Trial
Brief Title: Bring BPaL2Me Trial Comparing Nurse-Led RR-TB Treatment to Physician-Led RR-TB Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Witwatersrand, South Africa (Other); University of Cape Town (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB00234475; R01AI177135-01 (NIH)
Record Dates: First submitted 2022-12-20; First posted 2023-01-05 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Drug Resistant Tuberculosis
Keywords: nurse-led; non-inferiority cluster randomized trial; primary care; drug resistant tuberculosis; rifampicin resistant tuberculosis; human immunodeficiency virus; task sharing; South Africa
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Acquired Immunodeficiency Syndrome | interventions — Primary Health Care

STUDY DESIGN:
Intervention Model Description: Nurse-led primary care management for patients newly diagnosed with rifampicin-resistant tuberculosis (i.e. intervention) will be compared to physician-led, hospital-based management (i.e. standard of care)
Who Masked: Investigator, Outcomes Assessor
Masking Description: We will mask the investigators, statistician and safety review committee to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-Led Treatment in Primary Care (Experimental): At a primary care clinic intervention site, a nurse will be available once or twice weekly. The days/times will be dependent on clinic volume (i.e., cluster size), with scheduled rotations between PCCs. This rotation between PCC sites will mimic the physician's responsibilities/availability at a district hospital and creates parity between the trial arms. In this trial, we will have nurses dedicated to the management of RR-TB treatment, yet the volume at each site will not require the presence of a full-time nurse.
  Interventions: Other: Nurse-Led Treatment in Primary Care
- Physician-Led Treatment Hospital Based (No Intervention): Representing standard of care, primary care clinics will refer to hospital-based, physician-led care who will provide outpatient treatment. The typical clinical operations involve initiation of new patients once or twice weekly and PCCs are required to schedule a clinic day/time for the patient prior to referral (generally < 72 hours from the time of referral). All individuals receiving care at this site will receive care at the district RR-TB treatment program for the catchment area. For HIV co-infected persons, their HIV treatment is also transferred to the RR-TB physician with details about the HIV treatment communicated in the transfer of care letter. Physicians often cover multiple clinics and routinely take on call sessions on the weekend, due to staffing limitations, thus preventing their sole focus on the RR-TB program and limiting the number of days the RR-TB clinic offers new patient visits and, in most cases, days for follow-up visits.

INTERVENTIONS:
Other: Nurse-Led Treatment in Primary Care — At a primary care clinic intervention site, a nurse will be available once or twice weekly. The days/times will be dependent on clinic volume (i.e., cluster size), with scheduled rotations between PCCs. This rotation between PCC sites will mimic the physician's responsibilities/availability at a district hospital and creates parity between the trial arms. In this trial, we will have nurses dedicated to the management of RR-TB treatment, yet the volume at each site will not require the presence of a full-time nurse.
  Arms: Nurse-Led Treatment in Primary Care

SUMMARY:
The goal of the BringBPaL2Me Trial, a multi-principal investigator, multi-site, cluster randomized, non-inferiority trial is to compare nurse-led RR-TB treatment in primary care clinics to standard of care physician-led RR-TB treatment at district hospitals in the provinces of KwaZulu-Natal, Gauteng, and Eastern Cape.

The main aim is to conduct a 5-year, analyst and clinical safety review committee blinded, multi-site, cluster randomized trial to evaluate 1) treatment outcome; 2) safety; 3) patient associated catastrophic costs with the following hypotheses:

1. Outpatient nurse-led treatment in PCCs will be non-inferior to outpatient physician-led treatment at hospital-based outpatient sites among RR-TB patients, regardless of HIV co-infection, as determined by a successful treatment outcome [H1].
2. The proportion of SAEs identified will not significantly differ by blinded, independent review [H2].
3. Patient associated catastrophic costs (i.e., costs 20% or more of household income) will be lower in nurse-led treatment [H3].

DETAILED DESCRIPTION:
In South Africa (SA), nurses manage drug-susceptible Mycobacterium tuberculosis (TB) and TB/HIV coinfection within primary care clinics (PCCs); the TB treatment outcomes in this care model rival the best in the world. A primary care management strategy offers a convenient, patient-centered, model of care that integrates TB and HIV treatment within the same setting. However, a diagnosis of rifampicin-resistant TB (RR-TB), upends this model, requiring referral to a hospital-based, physician-led outpatient treatment center.

Hospital-based models add significant costs to patients, with estimates suggesting more than 80% of RR-TB patients experience catastrophic costs. Such added costs may decrease access to care, delay treatment receipt and contribute to loss to follow-up. One testable solution to this problem, however, is to move RR-TB care to primary care clinics led by nurses. The World Health Organization (WHO) released recommendations for RR-TB treatment earlier this year endorsing 6-month regimens and calling for decentralized, patient-centered models of care closer to the patient's home.

Although SA has long been a leading implementer of nurse-led models of care for TB and HIV due to large physician shortages and the National Department of Health's (NDoH) RR-TB Treatment Guidelines recommend integration of RR-TB within PCCs supporting both physician- and nurse-led models, utilization has been limited. While the team has spent the last decade building observational evidence around outcomes and safety, no randomized controlled trial evaluates nurse-led RR-TB treatment.

Secondary Aims: To evaluate clinical and cost-associated differentiators by arm:

1. Time to event analysis for a) RR-TB treatment initiation; b) smear/culture conversion; and, as applicable, c) HIV treatment initiation; d) HIV viral suppression; and e) AE and SAE symptom resolution.
2. Characterization of provider adherence to guidelines for: a) dosing requirements; b) RR-TB dosing changes based on AE and SAE events; and c) AE and SAE adjuvant medication management strategy.
3. Programmatic cost-effectiveness evaluation.

ELIGIBILITY:
Inclusion Criteria:

Cluster Inclusion Criteria:

Primary Care Clinics (PCCs) (i.e., clusters) are eligible if they meet the following:

1. within one of the selected hospital treatment catchment areas in Kwazulu-Natal, Gauteng and Eastern Cape Provinces;
2. willingness of provincial TB program managers and hospital leadership to participate;
3. willingness of PCC nurse manager to participate;
4. diagnosis of 10 or more RR-TB patients per year; and
5. have access to necessary labs, X-ray and electrocardiogram (ECG) equipment.

Participant Inclusion Criteria:

Adult participants aged 18 years of age and older, regardless of HIV status, who have a new RR-TB diagnosis, deemed willing and able to provide informed consent in one of the four most common SA languages [Zulu, Xhosa, Afrikaans, and English] will be eligible.

Participant Exclusion Criteria:

1. any clinical presentation requiring hospital admission or, in other words, the participant is not a candidate for outpatient primary care initiation (e.g., severe weakness, confusion, severe mental illness, symptomatic low blood pressure, severe shortness of breath, and temp >39.0);
2. Hemoglobin < 8mg/dL (from National Health Laboratory Service (NHLS) or point of care)) or liver disease (ALT > 120 U/L);
3. prolonged QTc>470ms, confirmed by 2 or more ecg;
4. rapid heartrate, tachycardia (HR >140); confirmed after 5 minutes of rest;
5. pregnancy;
6. evidence of extrapulmonary disease;
7. enrolled in another clinical trial that changes BPaL-L regimen, duration or symptom management process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2944 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
RR-TB treatment outcome | 6 months
  defined by the WHO will include the following: treatment success - the sum of cure and treatment completion; non-success - composite of each of the following negative outcomes: death, for any reason, while enrolled in RR-TB treatment (all-cause mortality); treatment failure - treatment terminated or need for permanent regimen change of at least two drugs because of: lack of culture conversion, bacterial reversion, worsening resistance profile, adverse events; and loss to follow-up interruption of 2 or more consecutive months of missed treatment.
Severe Adverse Events as assessed by the Division of AIDS (DAIDS) AE grading table | 12 months
  The following will be classified as an SAE using the DAIDS AE grading table for the purposes of this protocol:
  1. Lab abnormalities demonstrating grade 3 or higher: Myelosuppression (White blood cells (WBC), Red blood cells (RBC), Platelets); hepatotoxicity (Alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin); renal impairment (serum creatinine and creatinine clearance)
  2. Peripheral neuropathy, grade 3 or higher
  3. QT prolongation (Frederica's QTc), grade 3 or higher
  4. New onset seizure, regardless of grade
  5. Hospitalization, regardless of identified cause
  6. Mortality, regardless of identified cause
  7. All grade 4 AEs not listed above as an SAE
Patient associated catastrophic costs | 12 months
  (Costs 20% or more of household income) will be lower in nurse-led treatment

SECONDARY OUTCOMES:
Time to RR-TB treatment initiation | 60 days from trial screening
  Time to event analysis between diagnosis and treatment initiation
Time to smear/culture conversion | 120 days after treatment initiation
  Time to event analysis between treatment initiation and smear and culture conversion
Time to HIV treatment initiation | 120 days after treatment initiation
  Time to event analysis between enrollment and Antiretroviral therapy (ART) initiation
Time to HIV viral suppression | 6 months
  Time to event analysis between enrollment and HIV viral load < 200 copies
RR-TB dosing changes based on AE and SAE events | 12 months
  Provider appropriately manages RR-TB regimen based on AE and SAE events, as determined by blinded safety review
Time to adverse (AE) and severe (SAE) treatment related adverse event resolution | 12 months
  Time to event analysis for adverse and severe treatment related adverse events
Time to initiation of HIV prevention | 6 months
  Time to event analysis between enrollment and HIV prevention initiation for HIV negative patients
Provider adherence to dosing requirements, treatment initiation | 1 month
  Accuracy of regimen dosing based on treatment guidelines
AE and SAE adjuvant medication management strategy | 12 months
  Provider appropriately manages AE and SAE events, as determined by blinded safety review
Programmatic cost effectiveness evaluation | 12 months
  For the health system costs, we will use standard approaches outlined in "Value TB" costing guidelines for TB interventions. If the costs averted are found to be greater than the cost of the nurse-led PCC so that intervention saves money and is non-inferior, then it can be described as dominating (a more effective, less expensive choice) and it is economically the correct choice. In contrast, if the nurse-led PCC is non-inferior and yet more expensive, then we will calculate an incremental cost-effectiveness ratio (i.e., (CostNurse-CostUsual care)/(EffectNurse-EffectUsualCare)) that describes the extra costs necessary for each additional cured case.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Farley, PhD, MPH, ANP-BC, Principal Investigator — The Center for Infectious Disease and Nursing Innovation (CIDNI); Denise Evans, PhD, Principal Investigator — University of Witwatersrand, South Africa; Norbert Ndjeka, MBChB, Principal Investigator — University of Cape Town
Locations (5):
- South Africa (5):
  - Doris Goodwin Hospital, Pietermaritzburg, KwaZulu-Natal
  - Murchison Hospital, Port Shepstone, KwaZulu-Natal
  - King Dinuzulu TB Hospital, East London
  - Nkquebela TB Hospital, East London
  - Jose Pearson Hospital, Port Elizabeth

REFERENCES:
- [Background] van Rensburg C, Berhanu R, Hirasen K, Evans D, Rosen S, Long L. Cost outcome analysis of decentralized care for drug-resistant tuberculosis in Johannesburg, South Africa. PLoS One. 2019 Jun 6;14(6):e0217820. doi: 10.1371/journal.pone.0217820. eCollection 2019. PMID 31170207
- [Background] Laurence YV, Griffiths UK, Vassall A. Costs to Health Services and the Patient of Treating Tuberculosis: A Systematic Literature Review. Pharmacoeconomics. 2015 Sep;33(9):939-55. doi: 10.1007/s40273-015-0279-6. PMID 25939501
- [Background] Ho J, Byrne AL, Linh NN, Jaramillo E, Fox GJ. Decentralized care for multidrug-resistant tuberculosis: a systematic review and meta-analysis. Bull World Health Organ. 2017 Aug 1;95(8):584-593. doi: 10.2471/BLT.17.193375. PMID 28804170
- [Background] Masuku SD, Berhanu R, Van Rensburg C, Ndjeka N, Rosen S, Long L, Evans D, Nichols BE. Managing multidrug-resistant tuberculosis in South Africa: a budget impact analysis. Int J Tuberc Lung Dis. 2020 Apr 1;24(4):376-382. doi: 10.5588/ijtld.19.0409. PMID 32317060
- [Background] Crowley T, Mokoka E, Geyer N. Ten years of nurse-initiated antiretroviral treatment in South Africa: A narrative review of enablers and barriers. South Afr J HIV Med. 2021 Mar 11;22(1):1196. doi: 10.4102/sajhivmed.v22i1.1196. eCollection 2021. PMID 33824736
- [Background] Uebel KE, Fairall LR, van Rensburg DH, Mollentze WF, Bachmann MO, Lewin S, Zwarenstein M, Colvin CJ, Georgeu D, Mayers P, Faris GM, Lombard C, Bateman ED. Task shifting and integration of HIV care into primary care in South Africa: the development and content of the streamlining tasks and roles to expand treatment and care for HIV (STRETCH) intervention. Implement Sci. 2011 Aug 2;6:86. doi: 10.1186/1748-5908-6-86. PMID 21810242